CLINICAL TRIAL: NCT03431402
Title: Effects of Repetitive Hyperbaric Oxygen Therapy in Patients With Acute Ischaemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tamer Salah aldin Fahmy, Professor of critical care medicine, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KasrELAiniH critical care dep.
Record Dates: First submitted 2018-02-01; First posted 2018-02-13 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute stroke receive hyperbaric oxygen (Other)
  Interventions: Drug: Hyperbaric oxygen
- Acute stroke receive only conventional treatment (No Intervention)

INTERVENTIONS:
Drug: Hyperbaric oxygen — - HBOT group will receive 10 sessions of HBOT at 2.0 Atmosphere absolute (ATA) for one hour in a hyperbaric chamber pressured with compressed air, whereby patients will breath 100% oxygen to 2 ATA started within 3-5days after the onset of stoke plus conventional therapy as antiplatelets therapy, correction of hypovolaemia , hypoxia and adequate nutrition
  Arms: Acute stroke receive hyperbaric oxygen

SUMMARY:
Background and Rationale:

Cerebrovascular disease is always ranked at the top causes of death and most of hospitalized acute stroke patients have ischemic stroke [1].

Although the mortality rate of acute ischemic stroke is less than that of hemorrhagic stroke [1], it still results in patient disabilities and complications that often lead to significant costs to individuals, families, and society.

Traditional treatment for acute ischemic stroke includes thrombolytic therapy by injecting tissue plasminogen activator (t-PA) within three hours after onset of symptoms [2], antiplatelets and/or anticoagulant agents administered within the first 48 hours. Clinically, the narrow time window of thrombolytic therapy and coexisting contraindications limit the use of t-PA [2]. Thus, searching for an effective supplemental treatment for acute ischemic stroke is imperative.

Hyperbaric oxygen therapy (HBOT) is valuable in treating acute carbon monoxide poisoning [3,4], air or gas embolism [5], facilitating wound healing [6] and has been used as an adjuvant treatment for many neurological disorders that need further study as concussion [7] , stroke [8,9], cerebral palsy [ 10],traumatic brain injury [ 11], cerebral air embolism [12], Autism [13] and multiple sclerosis [14].

Indications of hyperbaric oxygen therapy recommended by undersea and hyperbaric medical society (UHMS) [15] are 1.air or gas embolism [5], 2.carbon monoxide poisoning [3,4], 3.clostridial myositis and myonecrosis [16], 4.crush injury, compartment syndrome and other acute traumatic ischemias [17], 5.decompression sickness [18], 6.arterial insufficiencies [19], 7.severe anemia [20], 8.intracranial abscess [21], 9.necrotizing soft tissue infections [22],10. refractory osteomyelitis [23], 11.delayed radiation injury [24], 12.compromised grafts and flaps [25], 13.acute thermal burn injury [26] and 14.idiopathic sudden sensorineural hearing loss [27].

Known mechanisms of HBOT-induced neuroprotection include enhancing neuronal viability via increased tissue oxygen delivery to the area of diminished blood flow, reducing brain edema, and improving metabolism after ischemia [28,29]. Furthermore, a recent study performed on a rat suggested that upregulation of the expression of glial derived neurotrophic factor (GDNF) and nerve growth factor (NGF) might underlie the effect of HBOT [30].

The effectiveness of use of Hyperbaric oxygen therapy in human ischemic stroke is still controversial that need further evaluation.

DETAILED DESCRIPTION:
Study Methods:

Study Population A 60 adult (aged >18 years) patients were included with a diagnosis of acute thromboembolic ischemic stroke within 48 hours after onset, according to clinical picture and imaging findings by brain computed tomography (CT) without evidence of hemorrhage, upon admission to the hospital and no patient received thrombolytic therapy.

Inclusion criteria:

Group one, HBOT group (n = 30): thirty adult patients with acute ischemic stroke will receive conventional medical treatment ( as antiplatelet but not thrombolytic therapy) with 10 sessions of adjunctive hyperbaric oxygen therapy (HBOT) within 3-5 days after the onset of stroke .

Compared with Group two, control group(n = 30): thirty adult patients with acute ischemic stroke will receive conventional medical treatment alone.

The baseline clinical characteristics were similar in both groups.

Exclusion criteria:

* Patient with cerebral hemorrhage
* Patient received thrombolytic therapy
* Emphysema with carbon dioxide retention
* Pneumothorax
* Seizure disorder
* Uncontrolled high fever

Demographic Characteristics:

Adults more than 18 years, Any gender. All patients upon admission to the hospital will provide:

Complete history taking:Age, Gender, Smoking, Alcohol consumption, Past history: diabetes mellitus , hypertension , Chronic obstructive pulmonary disease, Epilepsy or cardiovascular disease.

Neurological assessment use NIHSS score Blood tests:Complete blood count , Coagulation profile, Fasting blood sugar., Renal function test (Urea and creatinine).

CT brain

Chest x-ray :

Electrocardiogram (ECG):

ELIGIBILITY:
Inclusion criteria:

* Adult patients with acute ischemic stroke
* Glasgow coma scale more than 10

Exclusion criteria:

* Patient with cerebral hemorrhage
* Patient received thrombolytic therapy
* Emphysema with carbon dioxide (CO2) retention
* Pneumothorax
* Seizure disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in national institute of health stroke score before and after treatment with hyperbaric oxygen therapy | 2 years
  The national institute of health stroke score (NIHSS) is a 15 item neurologic examination that provides a quantitative measure of stroke-related neurologic deficit. (Maximum score of 42) "Mild" disease was defined as score of 0-14, "moderate" as 15-28, and "severe" as 29-42.
  As pretreatment evaluation, all patients will be evaluated by national institute of health stroke score within 48 hours after admission.
  As posttreatment evaluation, patients in the hyperbaric oxygen therapy group were evaluated by national institute of health stroke score after 10 sessions of hyperbaric oxygen therapy.
  The control group was evaluated with national institute of health stroke score 10 days after stroke onset.
  One month after treatment, all patients were evaluated again using the national institute of health stroke score.

SECONDARY OUTCOMES:
Hospital mortality | 2 years
Hospital length of stay | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim Shehata Hussin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes